CLINICAL TRIAL: NCT03000244
Title: Long-Term Follow up of Patients Undergoing Hematopoietic Stem Cell Transplantation
Brief Title: Long-Term Follow-up of People Undergoing Hematopoietic Stem Cell Transplantation
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170027; 17-C-0027
Record Dates: First submitted 2016-12-21; First posted 2016-12-22 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-11-18

CONDITIONS: Hematopoietic Stem Cell Transplantation; Tissue Donors
Keywords: Natural History; HCT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1/Patients: Patients who underwent hematopoietic stem cell transplant for any indication (malignant or non-malignant).
- 2/Donors: Related stem cell donors of those in Patients cohort.
- 3/Parents of patients: Parents/guardians of minors enrolled in cohort 1

SUMMARY:
Background:

People who have had an allogeneic hematopoietic stem cell transplant (HCT) have bone marrow or an immune system that is damaged. They get stem cells from a donor who is a relative. Researchers want to study stem cell donors and recipients to learn about the long-term effects of HCT. They want to learn how the stem cells change and how to improve their ability to fight cancer.

Objective:

To provide long-term follow-up care for people who underwent or will undergo HCT. To collect data, blood, and tissue samples to learn about late complications after HCT.

Eligibility:

Adults age 18 and older who will undergo HCT or underwent HCT and are surviving one year or more from the date of HCT. The stem cell donors for these recipients are also needed.

Design:

Recipients will have 1 visit each year. They will have a physical exam. They will answer questions about their medical history and health. They will receive screening and surveillance testing. They will complete brief questionnaires.

Recipients will have blood tests. They may have tissue biopsies or specimens (such as tissue in their cheek or skin or bone marrow biopsy).

Recipients will give their current address and phone number, and the same data for one or two other people, who can get in contact with them.

After the first visit at the clinic, some recipients may see a doctor close to home to get the necessary information and send it to NIH.

Donors will come to the clinic for 1 visit. They will answer questions about their medical history. Blood samples will be taken.

DETAILED DESCRIPTION:
Background:

* Patients who survive more than 3 years after allogeneic hematopoietic stem cell transplantation (HCT) have a high probability of being cured from their underlying disease; however, mortality rates remain 4 to 9-fold higher than the general population for at least 30 years after HCT.
* The most common causes of late mortality in HCT survivors include second malignancies, relapsed/recurrent disease, infections, chronic graft-versus-host disease (GVHD), respiratory diseases, and cardiovascular diseases.
* Guidelines for recommended screening and preventive practices for long-term survivors after HCT have been developed, and can be implemented to detect or prevent late complications after HCT.
* Understanding the pattern of immune reconstitution and immune dysregulation after HCT may help to elucidate the root mechanisms of late complications.

Objective:

-To collect clinical data on patients and late complications after HCT

Eligibility:

* Patients who underwent HCT for any indication and are surviving one year or more from the date of HCT
* Related stem cell donors of patients meeting the above criteria who participated or will be participating as a donor of stem cells or leukocytes.
* Age >= 4 years
* Any active disease relapse or new hematologic malignancy including post-transplant lymphoproliferative disorder (PTLD) are excluded from protocol enrollment.

Design:

* Prospective, longitudinal study of the natural history of long-term survivors after HCT.
* Clinical data on post-transplant complications and peripheral blood samples will be collected at yearly evaluations by the Principal Investigator, LAI, AI or representative investigator of the original HCT protocol.
* If patient develops complications such as new cancers, relapsed disease, new hematologic malignancy or PTLD they are exempt from required evaluations, and followed for survival and causes of death (management of complications as per primary team).
* As this is a longitudinal registry study without any planned intervention, there is no formal statistical analysis plan or accrual goal; descriptive data will be reported.

ELIGIBILITY:
* INCLUSION CRITERIA FOR PATIENT SUBJECTS:
* Patients who underwent HCT for any indication (malignant or non-malignant) and are surviving one year or more from the date of HCT (patients may be at any time point after HCT as long as it is >=1 year).
* Age >= 4 years
* Ability of patient or patient's Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document
* Patients will need to have a primary physician within the US (primary care, oncologist, hematologist, etc.) that will provide continued comprehensive care throughout the patient's participation in the study

EXCLUSION CRITERIA FOR PATIENT SUBJECTS:

-Patients with active disease relapse or new hematologic malignancy including post-transplant lymphoproliferative disorder (PTLD) are excluded from protocol enrollment.

INCLUSION CRITERIA FOR DONOR SUBJECTS:

* Related stem cell donors of patients meeting the above criteria as a donor of stem cells or leukocytes
* Age >= 4 years
* Ability of patient or patient's Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed

consent document

INCLUSION CRITERIA FOR PARENTS COMPLETING SURVEYS:

* Parents/guardians of minors enrolled on the study who have undergone HCT
* Willingness to complete surveys about the minor that underwent HCT

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have received an allogeneic stem cell transplant as well as donors of stem cells who are related to the patients who are study participants. Parents of minor recipients may also be enrolled to complete surveys. Participants can be from any community or co-enrolled on another NIH protocol.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-04-26 (Actual); Primary Completion 2050-08-12 (Estimated); Study Completion 2050-08-12 (Estimated)

PRIMARY OUTCOMES:
Basic characteristics of the patient population | at death
  Survival

SECONDARY OUTCOMES:
Provide a mechanism to ensure implementation of standard of care recommendations for post-transplant followup | Ongoing throughout study
  Observation of adherence and effects of standard of care recommendations
Obtain blood samples from stem cell transplant donors to study how biological factors related to the donor are associated with late complications | Ongoing throughout study
  Studying donor samples for potential correlations to transplant recipient complications.
Obtain blood and tissue samples to study and document immunologic reconstitution after stem cell transplant | Ongoing throughout study
  Immune monitoring for analysis
Monitoring of late effects after stem cell transplant for patients of ETIB protocols | Ongoing throughout study
  Survival and observation of long-term outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Najla El Jurdi, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared.@@@@@@All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Data from this study may be requested by contacting the PI.@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-C-0027.html